CLINICAL TRIAL: NCT06132672
Title: Identifying and Addressing Historical and Structural Drivers of Medical Mistrust Among Hispanic/Latino Gay, Bisexual and Other Men Who Have Sex With Men
Brief Title: Medical Mistrust Among Hispanic/Latino Gay, Bisexual and Other Men Who Have Sex With Men (HLMSM)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00101348; 1U01PS005250 (NIH)
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Human Immunodeficiency Virus
Keywords: Hispanic/Latino gay; bisexual men; HIV prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Recruit, enroll, and collect baseline data from 144 Hispanic/Latino Gay, Bisexual and Other Men Who Have Sex With Men (HLMSM), including 16 Community-Based Peer Navigators (known as Navigators) and their social network members (n=8 unique social network members per leader). Navigators (coupled with their social networks) will be randomly assigned to intervention (n=8 Navigators; n=64 social network members) or delayed-intervention (n=8 Navigators; n=64 social network members) groups. Navigators in the intervention group will be trained and supported for 12 months of implementation across years 3 and 4; those in the delayed-intervention group will be trained in year 5
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigators (peer navigator) training (Experimental): Training is designed to increase knowledge and skills. Navigators in the intervention group will be trained and supported for 12 months of implementation across years 3 and 4
  Interventions: Behavioral: Navigators (peer navigator) training
- delayed-intervention group (Experimental): Training is designed to increase knowledge and skills. The delayed-intervention group will be trained in year 5
  Interventions: Behavioral: delayed-intervention

INTERVENTIONS:
Behavioral: Navigators (peer navigator) training — The Navigators training will be designed to increase knowledge and skills to help others (i.e., social network members). Navigators in the intervention group will be trained and supported for 12 months of implementation across years 3 and 4
  Arms: Navigators (peer navigator) training
Behavioral: delayed-intervention — Those in the delayed-intervention group will be trained in year 5
  Arms: delayed-intervention group

SUMMARY:
There is an urgent need to address HIV inequities and disparities in the US, particularly within vulnerable communities such as Hispanic/Latino gay, bisexual, and other men who have sex with men (HLMSM).

DETAILED DESCRIPTION:
Medical mistrust is associated with HIV disparities among HLMSM because mistrust may result in delayed or reduced use of needed HIV prevention (e.g., HIV testing and Pre-exposure prophylaxis (PrEP) uptake) and care (e.g., AntiretroViral Therapy [ART]) services.

While advances have been made to increase the use of HIV prevention and care services, profound disparities persist, and a need remains for increased understanding of the multilevel drivers of medical mistrust and for effective interventions to address these drivers among HLMSM in the US.

This research proposes a mixed-method study that includes rigorous qualitative and quantitative methods to better understand the drivers of medical mistrust among Spanish-speaking, English-speaking, and bilingual (including Spanish and English, or an indigenous language and Spanish and/or English) HLMSM. This study also proposes to refine and test a multilevel intervention designed to address medical mistrust and increase the use of needed HIV prevention and care services among diverse HLMSM in Mecklenburg County, NC, a jurisdiction prioritized by the Ending the HIV Epidemic in the US (EHE) initiative.

ELIGIBILITY:
Inclusion Criteria:

* reside in Mecklenburg County, NC
* identify as Hispanic/Latino
* be ≥18 years of age
* speak English and Spanish
* report identifying as male and having had sex with at least 1 man in the past 6 months
* provide informed consent

Exclusion Criteria:

* less than 18 years of age
* female

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 144 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in Rate of medical mistrust | baseline to post-intervention up to 18 months
  The Group-Based Medical Mistrust Scale (GBMMS) - The response key was a Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree) and the score range was 12 to 60 - higher scores indicate greater levels of medical mistrust
Change in Rate of Human Immunodeficiency Virus (HIV) testing | baseline to post-intervention up to 18 months
  Change in Rate of Human Immunodeficiency Virus (HIV) testing - Self-Report - did participant use testing in past 12 months
Change in Rate of pre-exposure prophylaxis (PrEP) uptake | baseline to post-intervention up to 18 months
  Change in Rate of pre-exposure prophylaxis (PrEP) uptake - did participant use PrEP in past 12 months
Change in the amount of use of HIV care services | baseline to post-intervention up to 18 months
  Change in the amount of use of HIV care services - did participant use HIV care in past 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Rhodes, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing data generated from this study is an essential part of our proposed activities. This study will generate both quantitative and qualitative data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Last 6 months of Year 5
Access Criteria: De-identified data and associated documentation (including codebooks) will be available from the Principal Investigators under a data-sharing agreement with users that provides for a commitment to:
  (1) using the data for research purposes; (2) securing the data using appropriate computer technology; and (3) to destroying or returning the data after analyses are completed